CLINICAL TRIAL: NCT03875339
Title: Communities Helping the Hearing of Infants by Reaching Parents: The CHHIRP Navigator Trial
Brief Title: Communities Helping the Hearing of Infants by Reaching Parents
Acronym: CHHIRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matthew Bush, MD (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Matthew Bush, MD, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 47997 2019; 1R01DC017770-01 (NIH)
Record Dates: First submitted 2019-03-08; First posted 2019-03-14 (Actual); Results first posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Congenital Hearing Loss
Keywords: Infant Hearing Screening; Patient Navigator

STUDY DESIGN:
Intervention Model Description: Parallel Assignment via Stepped Wedge Trial Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Navigator Arm (Active Comparator): Examination of adherence to follow-up with a navigator.
  Interventions: Behavioral: Navigator Guidance
- Non-Intervention Arm (No Intervention): Examination of adherence to follow-up without a navigator.

INTERVENTIONS:
Behavioral: Navigator Guidance — Use of a dedicated Navigator to determine if follow-up and compliance rates can be improved for those infants initially demonstrating an abnormal hearing result.
  Arms: Navigator Arm

SUMMARY:
Hearing loss is the most common sensory congenital disorder and this condition is diagnosable and treatable. Children that are born with hearing loss have to undergo several hearing tests to diagnose the condition and many families are delayed in receiving this testing or never obtain the needed testing. This research employs a new method for helping children with hearing loss receive timely care by using a patient navigator, who is someone who teaches and provides emotional/social support for the families of these children.

The hypothesis of this study is that a patient navigator will hasten the timing of pediatric audiological testing, improve compliance with scheduled appointments, and expand parental knowledge of pediatric hearing loss.

DETAILED DESCRIPTION:
For Specific Arm 1:

The investigators will (1) use a stepped-wedge trial design to deliver patient navigation (PN) sequentially in 10 state-funded Kentucky Commission for Children with Special Healthcare Needs (CCSHCN) (also referred to as the Office for Children with Special Healthcare needs or OCSHCN) clinics randomized to cross from usual care to PN in steps of 6-month intervals over the project period. Prior to initiation of PN at each clinic, the control condition will be the standard of care. The overall effectiveness of PN will be tested by comparing non-adherence rates during the PN condition to those during the standard of care condition. Simultaneously, the investigators will (2) assess preliminary implementation outcomes (i.e., acceptability, adoption, recruitment/retention, and fidelity) as well as multilevel factors influencing implementation of PN in each clinic.

For Specific Arm 2:

Patient navigators will not be used for all subjects at participating clinics.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for parent-infant dyads:

1. Infant failed a hearing screening in one or both ears before postnatal hospital discharge
2. Infant was referred for follow-up diagnostic testing at one of the 10 participating CCSHCN clinics.
3. Parent able to speak either English or another language using Cyracom phone interpreting services.

Exclusion Criteria:

1. Children and parents live outside Kentucky or who will be moving out of Kentucky within the first three months of life.

Max Age: 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2699 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew L Bush, MD, PhD, Principal Investigator — Associate Professor, Vice Chair of Research
Locations (2):
- United States (2):
  - University of Kentucky, Lexington, Kentucky
  - Office for Children with Special Health Care Needs, Louisville, Kentucky

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made publicly available (by request to the PI) immediately following the acceptance for publication of the main findings from the final dataset.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: De-identified data will be made publicly available (by request to the PI) immediately following the acceptance for publication of the main findings from the final dataset.
Access Criteria: De-identified data will be made publicly available (by request to the PI) immediately following the acceptance for publication of the main findings from the final dataset.

REFERENCES:
- [Derived] Bush M, Hatfield M, Schuh M, Balasuriya B, Mahairas A, Jacobs J, Studts C, Westgate P, Schoenberg N, Shinn J, Creel L. Communities Helping the Hearing of Infants by Reaching Parents (CHHIRP) through patient navigation: a hybrid implementation effectiveness stepped wedge trial protocol. BMJ Open. 2022 Apr 19;12(4):e054548. doi: 10.1136/bmjopen-2021-054548. PMID 35440449

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first wave of the stepped-wedge intervention began in January 2020. In the original design, new clinics were supposed to launch every 6 months. Unfortunately, COVID shutdowns halted study activities, and the second wave was not launched until March 2021. The remaining waves occurred on a compressed timeline until the final clinic was launched in March of 2023. Once a clinic entered the intervention arm, they remained in the intervention condition until recruitment ended in September 2023.
Pre-assignment Details: While the study design describes "dyads" consisting of infants referred to testing and their parent/guardian, only the infants are considered participants because the outcome of the study describes the number of newborn infants who do not receive diagnostic audiological testing within 3 months of birth. Parents were not considered to be enrolled participants. Participants were counted only once, separate participants are included in each period below.
Units Other Than Participants: State-run healthcare clinics
Groups:
- Wave 1: Usual Care Months 1-6, Intervention Month 7 Onward: Wave 1: From month 1-6, one of the participating clinics delivered usual care to all patients referred for a follow-up hearing test. Beginning in Month 7, Patient Navigation became available for all participants referred to this clinic.
  The remaining 9 clinics deliver usual care until the intervention condition is activated during their "wave."
- Wave 2: Usual Care Months 1-20, Intervention Month 21 Onward: Wave 2: From month 1-20 two of the participating clinics delivered usual care to all patients referred for a follow-up hearing test. Beginning in Month 21, Patient Navigation became available for all participants referred to this clinic.
  The remaining 7 clinics deliver usual care until the intervention condition is activated during their "wave."
- Wave 3: Usual Care Months 1-25, Intervention Month 26 Onward: Wave 3: From month 1-25, two of the participating clinics delivered usual care to all patients referred for a follow-up hearing test. Beginning in Month 26, Patient Navigation became available for all participants referred to this clinic.
  The remaining 5 clinics deliver usual care until the intervention condition is activated during their "wave."
- Wave 4: Usual Care Months 1-31, Intervention Month 32 Onward: Wave 4: From month 1-31, two of the participating clinics delivered usual care to all patients referred for a follow-up hearing test. Beginning in Month 32, Patient Navigation became available for all participants referred to this clinic.
  The remaining 3 clinics deliver usual care until the intervention condition is activated during their "wave."
- Wave 5: Usual Care Months 1-32, Intervention Month 33 Onward: Wave 5: From month 1-32 one of the participating clinics delivered usual care to all patients referred for a follow-up hearing test. Beginning in Month 33, Patient Navigation became available for all participants referred to this clinic.
  The remaining 2 clinics deliver usual care until the intervention condition is activated during their "wave."
- Wave 6: Usual Care Months 1-37, Intervention Month 38 Onward: Wave 6: From month 1-37 one of the participating clinics delivered usual care to all patients referred for a follow-up hearing test. Beginning in Month 38, Patient Navigation became available for all participants referred to this clinic.
  The remaining 1 clinic delivers usual care until the intervention condition is activated during their "wave."
- Wave 7: Usual Care Months 1-44, Intervention Month 45: Wave 7: From month 1-44 one of the participating clinics delivered usual care to all patients referred for a follow-up hearing test. Beginning in Month 45, Patient Navigation became available for all participants referred to this clinic.
  No clinics remain in the "usual care condition" at Month 45.
Period: Usual Care
Arm/Group | Wave 1: Usual Care Months 1-6, Intervention Month 7 Onward | Wave 2: Usual Care Months 1-20, Intervention Month 21 Onward | Wave 3: Usual Care Months 1-25, Intervention Month 26 Onward | Wave 4: Usual Care Months 1-31, Intervention Month 32 Onward | Wave 5: Usual Care Months 1-32, Intervention Month 33 Onward | Wave 6: Usual Care Months 1-37, Intervention Month 38 Onward | Wave 7: Usual Care Months 1-44, Intervention Month 45
Started | 452; 1 State-run healthcare clinics | 278; 2 State-run healthcare clinics | 235; 2 State-run healthcare clinics | 31; 2 State-run healthcare clinics | 45; 1 State-run healthcare clinics | 31; 1 State-run healthcare clinics | 26; 1 State-run healthcare clinics
Completed | 452; 1 State-run healthcare clinics | 278; 2 State-run healthcare clinics | 235; 2 State-run healthcare clinics | 31; 2 State-run healthcare clinics | 45; 1 State-run healthcare clinics | 31; 1 State-run healthcare clinics | 26; 1 State-run healthcare clinics
Not Completed | 0; 0 State-run healthcare clinics | 0; 0 State-run healthcare clinics | 0; 0 State-run healthcare clinics | 0; 0 State-run healthcare clinics | 0; 0 State-run healthcare clinics | 0; 0 State-run healthcare clinics | 0; 0 State-run healthcare clinics
Period: Patient Navigation Available
Arm/Group | Wave 1: Usual Care Months 1-6, Intervention Month 7 Onward | Wave 2: Usual Care Months 1-20, Intervention Month 21 Onward | Wave 3: Usual Care Months 1-25, Intervention Month 26 Onward | Wave 4: Usual Care Months 1-31, Intervention Month 32 Onward | Wave 5: Usual Care Months 1-32, Intervention Month 33 Onward | Wave 6: Usual Care Months 1-37, Intervention Month 38 Onward | Wave 7: Usual Care Months 1-44, Intervention Month 45
Started | 36; 1 State-run healthcare clinics | 795; 2 State-run healthcare clinics | 283; 2 State-run healthcare clinics | 342; 2 State-run healthcare clinics | 97; 1 State-run healthcare clinics | 21; 1 State-run healthcare clinics | 27; 1 State-run healthcare clinics
Completed | 36; 1 State-run healthcare clinics | 795; 2 State-run healthcare clinics | 283; 2 State-run healthcare clinics | 342; 2 State-run healthcare clinics | 97; 1 State-run healthcare clinics | 21; 1 State-run healthcare clinics | 27; 1 State-run healthcare clinics
Not Completed | 0; 0 State-run healthcare clinics | 0; 0 State-run healthcare clinics | 0; 0 State-run healthcare clinics | 0; 0 State-run healthcare clinics | 0; 0 State-run healthcare clinics | 0; 0 State-run healthcare clinics | 0; 0 State-run healthcare clinics

BASELINE CHARACTERISTICS:
Population: Infants referred to state-run clinics for follow-up testing after a failed newborn hearing screening.
Groups:
- Total: Total of all reporting groups
Arm/Group | Navigator Arm | Non-Intervention Arm | Total
Number analyzed (Participants) | 1601 | 1098 | 2699
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1601 | 1098 | 2699
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 712 | 455 | 1167
  Male | 889 | 643 | 1532
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1601 | 1098 | 2699

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who do Not Receive Diagnostic Audiological Testing (Aim 1)
Description: This outcome is the number of participants who do not follow-up at an OCSHCN Clinic for diagnostic audiologic testing after a failed newborn hearing screening from the date of randomization to 3 months after birth.
Time Frame: 3 months. (This is the amount of time from an abnormal screen at birth to an expected follow-up at a clinic or hospital.)
Measure: Count of Participants; unit: Participants
Arm/Group | Navigator Arm | Non-Intervention Arm
Number analyzed (Participants) | 1601 | 1098
Participants | 378 | 336

ADVERSE EVENTS:
Time Frame: Nine months.
Description: Parents were not considered enrolled, adverse event data reported is for infants only.
Arm/Group | Navigator Arm | Non-Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/1601 | 0/1098
Serious Adverse Events (participants affected / at risk) | 0/1601 | 0/1098
Other Adverse Events (participants affected / at risk) | 0/1601 | 0/1098

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-04): https://cdn.clinicaltrials.gov/large-docs/39/NCT03875339/Prot_SAP_001.pdf
  • Informed Consent Form (2023-04-08): https://cdn.clinicaltrials.gov/large-docs/39/NCT03875339/ICF_000.pdf